CLINICAL TRIAL: NCT03584295
Title: A Multicentre, Randomized-controlled Trial of EXtracorporeal CO2 Removal to Facilitate Early Extubation Compared to Invasive Mechanical Ventilation in Patients with Severe Acute Exacerbation of COPD (X-COPD)
Brief Title: Early Extubation by ECCO2R Compared to IMV in Patients with Severe Acute Exacerbation of COPD
Acronym: X-COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Xenios AG (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Organization: Fresenius Medical Care Deutschland GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPD-ECCO2R-01-INT
Record Dates: First submitted 2018-06-25; First posted 2018-07-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional care (Active Comparator): Patients with acute exacerbation of severe COPD, requiring invasive mechanical ventilation treated with Conventional care. Conventional care includes invasive mechanical ventilation and the attempt to extubate the patient and switch to NIV. If extubation fails tracheostomy can be performed according to the treating physician.
  Interventions: Other: Conventional Care
- Extracorporeal carbon dioxide removal (Experimental): Patients with acute exacerbation of severe COPD, requiring invasive mechanical ventilation will be treated with vv-ECCO2R (Extracorporeal carbon dioxide removal) to facilitate early extubation. ECCO2R is used in a standard configuration with either double lumen cannula (22-24Fr) or two small single vessel cannulas (15-19 Fr), allowing a blood flow rate between 1-1.75 L/min.
  Interventions: Device: Extracorporeal carbon dioxide removal

INTERVENTIONS:
Device: Extracorporeal carbon dioxide removal — Patients with acute exacerbation of severe COPD, requiring invasive mechanical ventilation will be treated with vv-ECCO2R to facilitate early extubation
  Arms: Extracorporeal carbon dioxide removal
Other: Conventional Care — Patient with acute exacerbation of severe COPD, requiring invasive mechanical ventilation treated with Conventional Care. Conventional care includes invasive mechanical ventilation and the attempt to extubate the patient and switch to NIV. If extubation fails tracheostomy can be performed according to the treating physician.
  Arms: Conventional care

SUMMARY:
The study aims to investigate if veno-venous (vv)-extracorporeal carbon dioxide Removal (ECCO2R) is capable of reducing mortality and/or severe disability at day 60 after randomisation in patients with severe acute exacerbation of chronic obstructive pulmonary disease (COPD) requiring invasive mechanical ventilation (IMV). Extubation will be facilitated by VV-ECCO2R and compared to IMV alone in a randomized controlled trial.

DETAILED DESCRIPTION:
The current study hypothesizes an advantage for veno-venous extracorporeal carbon dioxide removal (VV-ECCO2R) in severe acute exacerbation of COPD requiring invasive mechanical ventilation (IMV) to facilitate early extubation in terms of reducing mortality or severe disability. The study hypothesizes that avoiding IMV could reduce mortality and substantially improve quality of life, especially in regard to avoidance of tracheostomy and long-term home IMV. Improvement in mobility due to sooner recovery has a further major impact on patients' QoL.

After randomization patients with acute exacerbation of severe COPD, requiring invasive mechanical ventilation will be treated either with conventional care or VV-ECCO2R to facilitate early extubation. VV-ECCO2R is used in a standard configuration with either double lumen cannula (22-24Fr) or two small single vessel cannulas (15-19 Fr), allowing a blood flow rate between 1-1.75 L/min.

Conventional care in the control arm includes invasive mechanical ventilation and the attempt to extubate the patient as early as possible and to switch to non-invasive ventilation (NIV). If extubation fails, tracheostomy can be performed according to the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed and dated by the investigator; and

   1. if patient is able to give consent: by the study patient
   2. if patients unable to give consent: by the legal representative or
   3. if an emergency situation is determined: by an independent consultant physician.
2. Minimum age of 18 years
3. In case of female patients:

   1. Postmenopausal status defined as I. Prior bilateral oophorectomy Or II. Age ≥60 years Or if Age is <60 years or cannot be determined
   2. A negative pregnancy test, defined as negative beta hCG test with a hCG level <5 mIU/mL.
4. Known History of COPD
5. Acute exacerbation of COPD requiring invasive mechanical ventilation
6. Failed extubation attempt or extubation not possible within 24 hours after intubation
7. Acute and potentially reversible cause of respiratory failure as determined by the treating physician

Exclusion Criteria:

1. Any conditions which could interfere with the patient's ability to comply with the study
2. In case of female patients: pregnancy and lactation period
3. Participation in any interventional clinical study during the preceding 30 days
4. Platelets <70.000/µl at baseline
5. Previous participation in the X-COPD study
6. Endotracheally intubated and mechanically ventilated for >96 hours prior to randomization
7. Acute liver failure, defined by an international normalized ratio (INR) >2 without anticoagulation and/or bilirubin >4 mg/dL (>68 μmol/L) and/or hepatic encephalopathy (all three apply)
8. PaO2/FiO2 ratio <120 mmHg measured with FiO2 of 1.0
9. Expectation of disease progression leading to high-flow extracorporeal membrane oxygenation (ECMO) treatment
10. Cerebral haemorrhage
11. Tracheostomy
12. Estimated life expectancy <6 months due to reasons other than COPD
13. Acute ischemic stroke
14. Contraindication to anticoagulation
15. Severe chronic liver disease (Child Pugh C)
16. Acute pulmonary embolism requiring thrombolytic therapy
17. Acute or chronic heart failure with left ventricular ejection fraction <30%
18. Acute or chronic renal failure requiring dialysis
19. Organ transplantation or immunosuppression due to ongoing immunosuppressive medication or neutropenia for instance following organ transplantation or anticancer therapy
20. Neuromuscular disorder or chronic restrictive lung disease affecting native lung ventilation
21. Known Heparin induced thrombocytopenia type II
22. Acute coronary syndrome and myocardial infarction
23. Obesity hypoventilation syndrome
24. BMI >40
25. Patient not expected to survive 48 hours
26. Do not resuscitate (DNR) order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Death or severe disability | day 60
  Death or severe disability at day 60 after randomization, with severe disability defined as confinement to bed and/or inability to wash or dress alone and/or need for long-term invasive mechanical ventilation by day 60

SECONDARY OUTCOMES:
Mortality or severe disability at day 180 after randomization | Day 180
  Change in mortality/severe disability rate
Ventilator-associated pneumonia during ICU treatment | up to 60 days
  1. Some sign of respiratory distress, e.g., increased RR, increased FiO2
  2. New or enlarging infiltrates on CXR
  3. Culture of relevant organism from lung or major change in secretions from lung
Reintubation rate | until day 180 after randomization
  Number of reintubations
Days on IMV or noninvasive ventilation (NIV) or ECCO2R | up to 60 days
  defined as duration of total ventilatory support
Thrombosis during treatment period | up to 29 Days
  Thrombosis of major venous vessels during the treatment period
Quality of life of patient | up to 180 days
  Measured at day 60 and 180 after randomization, measured with Severe Respiratory Insufficiency and EQ-5D-5L Questionnaire
Renal function | up to 29 days
  Worsening of renal function
Mobility, measured with ActiGraph | up to 180 days
  Subgroup: Activity measurement with ActiGraph (at 1 centre)
Treatment Cost | up to 180 days
  Total Treatment costs for the hospital stay
Length of hospital stay | Up to 180 Days
  Change in days of hospital stay
Need of tracheostomy | Up to 180 Days
  Change in rate of tracheostomy
Breathing | up to 60 days
  Breathing through tracheostomy at day 60 after randomization
Readmission | Up to 180 Days
  Readmission to hospital within 180 days after randomization
Exacerbations | Up to 180 Days
  Number of exacerbations within 180 days after randomization
Severe Bleeding | up to 60 days
  Defined as any bleeding event requiring administration of 1 unit of packed red cells, Detection of severe bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Christian Karagiannidis, Prof. Dr., Principal Investigator — Kliniken der Stadt Köln gGmbH, ARDS and ECMO Zentrum Köln-Merheim
Locations (1):
- Kliniken der Stadt Köln gGmbH, ARDS and ECMO Zentrum Köln-Merheim, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No